CLINICAL TRIAL: NCT04866329
Title: FERTilité féminine, Agents ENvironnementaux et Stress OXydant
Brief Title: Female Fertility, Environmental Agents and Stress Oxidant
Acronym: FERTENOX
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR200209; 2020-A03241-38 (Other: IdRCB)
Record Dates: First submitted 2021-03-23; First posted 2021-04-29 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Female Infertility
Keywords: Environmental pollutants; Bisphenols; Ethynylestradiol; Glyphosate; Oxidative stress; Oocyte and embryo quality; In vitro fertilization; Pregnancy; Follicular fluid and urine biomarkers
MeSH Terms: conditions — Infertility, Female | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In Vitro Fertilisation protocol: Women followed in the department for an in vitro fertilisation protocol
  Interventions: Other: Blood sample; Other: Urine sample; Other: Follicular fluid and granulosa cells sample

INTERVENTIONS:
Other: Blood sample — Additional blood sampling at the end of ovarian stimulation monitoring (the eve of the oocyte pick-up)
Other: Urine sample — Collection of the first urine in the morning on the day of the oocyte pick-up
Other: Follicular fluid and granulosa cells sample — Collection of follicular fluid and granulosa cells during oocyte pick-up.

SUMMARY:
Synthetic products used in industrial, pharmaceutical, agro-alimentary or agricultural fields are found in our environment. Thus, humans could be simultaneously exposed to several of these pollutants. Furthermore, these environmental agents exert or could exert adverse actions on fertility, by altering gamete and embryo quality through endocrine disruptor effects or through increase in oxidative stress in gonads (cellular pathway known to be involved in several human reproductive pathologies).

In this context, the objectives of the present project are to obtain descriptive and analytical data on woman and oocyte exposure to several environmental agents (bisphenols, ethynylestradiol and glyphosate). The relation between these pollutant measures in follicular fluid and urine (from women receiving follow-up of in vitro fertilization (IVF) protocol in the University hospital of Tours, France) and the oocyte quality, the IVF and pregnancy successes will be studied. Several oxidative stress biomarkers in blood and follicular fluid will be also measured for these women, who will complete a questionnaire on their lifestyles. Finally, thanks to in vitro approaches, the effects and the mechanisms of action (including oxidative stress) of these pollutants (alone or in cocktails) will be studied on granulosa cells from these patients.

DETAILED DESCRIPTION:
After being informed about the project Fertenox during a meeting describing about the Fecondation In Vitro protocol, all women patients not opposing to participate in the study and to use individual information will be included in the research during the usual bacteriological exam performed 1-2 months before oocyte pick up in the University hospital. They will receive the questionnaire on their lifestyle during this exam.

On the eve of the oocyte pick up (at the end of ovarian stimulation) during the usual blood collection, three additional tubes of blood will be collected for each patient in the University hospital. Women will also receive the screw-top container for morning-after urine sample and the completion of the lifestyle questionnaire will be checked (some advices will be done if necessary to help patients to fill out the questionnaire). Samples will be treated, aliquoted and stored according to requirements the same day.

The day of the oocyte pick up, the first morning urine will be collected by patients at home (or otherwise in the hospital). The completed questionnaire will be recovered and follicular fluid and granulosa cells will be collected for each woman. Samples will be aliquoted and stored according to requirements the same day. Granulosa cells will be cultured for in vitro approaches in research labs the same day.

Tubes of blood, urine and follicular fluid will be coded and kept at -80°C in the University hospital until their shipment to laboratories, where analyses of pollutants (bisphenols, ethynylestradiol and glyphosate) and analyses of oxidative stress biomarkers (antioxidant vitamins, FRAP), activity of several enzymes (catalase, superoxide dismutase, glutathione peroxidase) and oxidized lipids) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 to 43 years old
* First oocyte puncture (IVF rank = 1)

Exclusion Criteria:

* Opposition to data processing
* IVF rank equal or greater than 2
* Egg donation
* Intracytoplasmic Sperm Injection with testicular biopsy
* Intracytoplasmic Sperm Injection with self-preservation straw
* Sperm donation

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women followed in the department for an in vitro fertilisation procedure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-12-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of ethinylestradiol in follicular fluid | Baseline
  Assessed by measure of ethinylestradiol in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Presence or absence of ethinylestradiol in urine | Baseline
  Assessed by measure of ethinylestradiol in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Presence or absence of bisphenols in follicular fluid | Baseline
  Assessed by measure of bisphenols in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Presence or absence of bisphenols in urine | Baseline
  Assessed by measure of bisphenols in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Presence or absence of glyphosate in follicular fluid | baseline
  Assessed by measure of glyphosate in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Presence or absence of glyphosate in urine | baseline
  Assessed by measure of glyphosate in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of ethinylestradiol in follicular fluid | baseline
  Assessed by concentration of ethinylestradiol in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of ethinylestradiol in urine | baseline
  Assessed by concentration of ethinylestradiol in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of bisphenols in follicular fluid | baseline
  Assessed by concentration of bisphenols in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of bisphenols in urine | baseline
  Assessed by concentration of bisphenols in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of glyphosate in follicular fluid | baseline
  Assessed by concentration of glyphosate in follicular fluid by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Concentration of glyphosate in urine | baseline
  Assessed by concentration of glyphosate in urine by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)

SECONDARY OUTCOMES:
Oocyte quality | baseline
  Assessed by nuclear maturity of each collected punctured oocyte
Embryo quality | Day 2 and day 5/6 after oocyte pick up
  Assessed by in vitro early embryo developmental competence of each punctured oocyte (Day 2 embryo morphology, ability to reach the blastocyst stage, Day 5/6 blastocyst morphology, blastocyst outcome (transfer, freezing, discarding)
Embryo implantation success (pregnancy success) | From day 7 after embryo transfer for beta hCG assay, at 8 weeks of amenorrhea for foetus cardiac activity and after birth
  Assessed by confirmation of a clinical pregnancy (blood beta human chorionic gonadotropin assay: > 1000 Unity Intenational /L), by confirmation of on-going pregnancy (ultrasound measure of foetus cardiac activity) and by confirmation delivery of live and healthy birth
Oxidative stress biomarkers in follicular fluid | baseline
  Assessed by measure of antioxidant vitamins (carotenoids, vitamin E, retinol) by High Performance Liquid Chromatography
Oxidative stress biomarkers in follicular fluid | Baseline
  Assessed by measure of oxidized lipids (isoprostanoids) by LC-MS/MS
Oxidative stress biomarkers in follicular fluid | Baseline
  Assessed by measure of antioxidant power (FRAP: Ferric ion Reducing Antioxidant Power) by spectrophotometry
Oxidative stress biomarkers in follicular fluid | Baseline
  Assessed by measure of glutathione peroxidase activity by spectrophometry
Oxidative stress biomarkers in blood | On the eve of baseline
  Assessed by measure of plasma antioxidant vitamins (carotenoids, vitamin E, retinol) by HPLC
Oxidative stress biomarkers in blood | On the eve of baseline
  Assessed by measure of plasma oxidized lipids (isoprostanoids) by LC-MS/M
Oxidative stress biomarkers in blood | On the eve of baseline
  Assessed by measure of plasma antioxidant power (FRAP) by spectrophotometry
Oxidative stress biomarkers in blood | On the eve of baseline
  Assessed by measure of activities of glutathione peroxidase, catalase and superoxide dismutase in red blood cells by UV and visible spectrophometry
Oxidative stress biomarkers in urine | baseline
  Assessed by measure of oxidized lipids (isoprostanoids) by LC-MS/MS
Information on woman lifestyles | The 3 last months of lifestyles before baseline
  Assessed by a questionnaire on sociodemographic characteristics, smoking, physical activity, professional and environmental expositions, consumption of dietary supplements (antioxidants), consumption of drinks (tap water, from plastic bottle, cans...), food reheating habit, consumption of food from tin box, use of hygiene and cosmetic products...
Pollutant effects on patient granulosa cells in vitro | after 24 or 48h of exposure
  Assessed on cellular viability (CCK8, live-dead assay)
Pollutant effects on patient granulosa cells in vitro | after 24 or 48h of exposure
  Assessed on proliferation (BrdU)
Pollutant effects on patient granulosa cells in vitro | after 48 or 72h of exposure
  Assessed on steroid production (ELISA, LC-MS)
Pollutant effects on patient granulosa cells in vitro | after 1 or 24h of exposure
  Assessed on energetic metabolism (mitochondrial and glycolytic activities by Seahorse and Omnilog assays)
Pollutant effects on patient granulosa cells in vitro | after 5, 6 or 24h of exposure
  Assessed on oxidative stress biomarkers (reactive oxygen production, Nrf2 nuclear translocation by confocal microscopy, cytometry and fluorimetry)
Pollutant effects on patient granulosa cells in vitro | after 24, 48 or 72h of exposure
  Assessed on protein expression (Western Blotting) of several markers of the studied functions (including oxidative stress)
Pollutant effects on patient granulosa cells in vitro | after 6 or 24h of exposure
  Assessed on gene expression (RNAseq and Quantitative Reverse Transcription-PCR) of several markers of the studied functions (including oxidative stress)
Pollutant effects on patient granulosa cells in vitro | after 1, 5, 10, 30 and 60 min of exposure
  Assessed on protein expression (Western Blotting ) of signaling pathways
Pollutant effects on patient granulosa cells in vitro | after 6h of exposure
  Assessed on gene expression (RNAseq and qRT-PCR) of signaling pathways

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice GUERIF, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Department of Reproductive Medicine and Biology, Univesity Hospital, Tours, Tours, France